CLINICAL TRIAL: NCT06191991
Title: A Phase 1 Study in Healthy Volunteers to Evaluate the Drug-Drug Interaction Potential Between ALG-055009 and Statin Therapy(Ies)
Brief Title: A Phase 1 Study to Evaluate the Drug-Drug Interaction Potential Between ALG-055009 and Statin Therapy(Ies)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aligos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ALG-055009-302
Record Dates: First submitted 2023-11-03; First posted 2024-01-05 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atorvastatin with ALG-055009 (Experimental): Single dose PO administration of 40 mg atorvastatin (Day 1), then a washout period of at least 2 days, followed by PO QD administration of 0.9 mg ALG-055009 for 14 days (Days 3-16) and single dose PO administration of 40 mg atorvastatin (Day 15).
  Interventions: Drug: Atorvastatin; Drug: ALG-055009
- Rosuvastatin with ALG-055009 (optional) (Experimental): Single dose PO administration of 10 mg rosuvastatin (Day 1), then a washout period of at least 4 days, followed by PO QD administration of 0.9 mg ALG-055009 for 11 days (Days 5-15) and single dose PO administration of 10 mg rosuvastatin (Day 11).
  Interventions: Drug: ALG-055009; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Atorvastatin — 40 mg
  Arms: Atorvastatin with ALG-055009
Drug: ALG-055009 — 0.9 mg
Drug: Rosuvastatin — 10 mg
  Arms: Rosuvastatin with ALG-055009 (optional)

SUMMARY:
This Phase 1 study consists of two parts, all conducted in healthy volunteers (HVs). In Parts 1 and 2, the drug-drug interaction (DDI) potential of ALG-055009 will be explored, where subjects will be assigned to receive multiple doses of ALG-055009 and 2 single doses of one of the following concomitant drugs: atorvastatin (Part 1), or rosuvastatin (Part 2, optional).

ELIGIBILITY:
Inclusion Criteria:

1. Subject must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study.
2. In the Investigator's opinion, the subject is able to understand and comply with protocol requirements, instructions, and protocol stated restrictions and is likely to complete the study as planned.
3. Male or female between 18 and 65 years of age, extremes included.
4. Female subjects must not be a woman of childbearing potential defined as:

   1. Postmenopausal:

      A postmenopausal state is defined as no menses for at least 12 months without an alternative medical explanation, confirmed by a high follicle-stimulating hormone (FSH) level in the postmenopausal range at screening.

      OR
   2. Permanently sterile:

   Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.
5. Male subjects must agree to wear a condom during sexual intercourse and their female sexual partners should agree to use effective means of contraception (Section 7.2.3). These contraceptive measures must be implemented, at a minimum, from the start of dosing until at least 90 days after the last dose.

   NOTE: Contraceptive use should be consistent with local regulations regarding the use of contraceptive methods for subjects participating in clinical studies.
6. Subjects must have a body mass index (BMI) of 18.0 to 32.0 kg/m2, extremes included.
7. Subjects must be nonsmokers for at least 3 months prior to enrollment.
8. Subjects must have a 12-lead electrocardiogram (ECG) that meets the following criteria at screening:

   1. Heart rate between 40 and 100 beats per minute [bpm], extremes included;
   2. QT interval corrected for heart rate (QTc) according to Fridericia's formula (QTcF) <450 ms (males) or <470 ms (females);
   3. QRS interval <120 ms;
   4. PR interval ≥110 to ≤220 ms;
   5. In addition to fulfilling the above ECG criteria, ECG morphology must have no clinically significant abnormalities observed.
9. Subjects must be deemed to be in good overall health by the Investigator on the basis of a medical evaluation that reveals the absence of any clinically significant abnormality and includes a physical examination, medical history, vital signs, and the results of blood chemistry, blood coagulation and hematology tests, and a urinalysis performed at screening.
10. Subject must be willing and able to adhere to the Prohibited Medication requirements (Appendix B) and Special Precautions (Section 6.12).

Exclusion Criteria:

1. Subject with a) a medical history of thyroid disorder or b) abnormal thyroid stimulating hormone (TSH), free thyroxine (T4) or total triiodothyronine (T3) during screening, and Day -1 or c) known sensitivity to thyroid medications.
2. The following laboratory values at screening are exclusionary:

   1. ALT or AST > upper limit of normal (ULN),
   2. Total bilirubin >1.2× ULN, unless Gilbert's Syndrome is suspected
3. Subjects with any current or previous illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject or that could prevent, limit, or confound the protocol specified assessments or study results' interpretation. This may include, but is not limited to, renal, cardiac, vascular, pulmonary, gastrointestinal, hepatologic, endocrine, neurologic, dermatologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances.
4. Subjects with a past history of cardiac arrhythmias, risk factors for Torsade de Pointes syndrome (e.g., hypokalemia, family history of long QT Syndrome) or history or clinical evidence at screening of significant or unstable cardiac disease such as: angina, congestive heart failure, myocardial infarction, diastolic dysfunction, significant arrhythmia, coronary heart disease, clinically significant ECG abnormalities, moderate to severe valvular disease or uncontrolled hypertension. Evidence on ECG of heart block or bundle branch block, inclusive of first-degree AV block and incomplete bundle branch block, is also exclusionary.
5. History of unexplained syncope.
6. Subjects with a history of clinically significant (in the opinion of the Investigator) drug allergy such as, but not limited to, sulfonamides or drug allergy witnessed in previous studies with experimental drugs.
7. Subjects with a recent (within 1 year of enrollment) history or current evidence of use of amphetamines, barbiturates, narcotic or other drugs of abuse/recreational drug use (including cannabis).
8. Excessive use of alcohol defined as regular consumption of ≥14 standard drinks/week for women and ≥21 standard drinks/week for men (Chalasani et al. 2018). For current definition of a standard drink, please refer to the National Institute on Alcohol Abuse and Alcoholism website (https://www.niaaa.nih.gov/what-standard-drink).
9. Unwilling to abstain from alcohol use for 1 week prior to start of study through end of study follow up.
10. Positive results for urine drug screen, alcohol or cotinine test at screening and Day -1.
11. Subjects with current:

    1. Hepatitis A virus infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]).
    2. Hepatitis B infection defined as presence of HBsAg or HBV core antibody.
    3. Hepatitis C virus (HCV) infection (confirmed by HCV antibody and/or HCV RNA).
    4. Hepatitis E virus: Anti-HEV IgM-positive and/or detectable HEV RNA level.
    5. Human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection (confirmed by antibodies) at screening.
    6. Acute infection at the time of enrollment. If an acute infection is considered resolved prior to enrollment, the subject remains eligible.
12. Male subjects who plan to father a child while enrolled in this study or within 90 days after the last dose of study drug.
13. Subject receiving, or urgently requiring, any lipid lowering therapy (e.g., statins). Prior use (at least 1 month prior to screening) of lipid lowering therapy is not exclusionary.
14. Subject who has taken or requires treatment with any disallowed therapies as noted in Prohibited Medications (Appendix B) and Special Precautions (Section 6.12) within 1 week or 5 half-lives (whichever is longer) before the planned first dose of study drug or during dosing; use of sensitive CYP3A4 substrates, inhibitors/inducers of CYP3A4, inhibitors of OATP1B1, OATP1B3, and/or BCRP transporters (see Appendix B), within 28 days or 5 half-lives (whichever is longer) prior to the first dose of study drug is prohibited.
15. Consumption of grapefruit, grapefruit juice, and Seville oranges within 14 days prior to study drug administration.
16. Consumption of apple or orange juice, citrus fruits, vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard), and charbroiled meats within 7 days prior to study drug administration.
17. Consumption of any food or drink/beverage containing quinine (e.g., tonic, bitter lemon, bitter alcoholic beverages containing quinine) within 24 hours prior to study drug administration.
18. Consumption of any food or drink/beverage containing poppy seeds or codeine containing formulation within 72 hours of screening and admission to study site.
19. Known hypersensitivity or previous adverse events (AEs) with atorvastatin, rosuvastatin or other statins.
20. Subjects who received an investigational agent within 4 weeks (or 5 half-lives, whichever is longer) prior to enrollment.
21. Subjects currently participating in another clinical or medical interventional research study.
22. Subjects with any laboratory result that is considered clinically significant by the Investigator at screening. Abnormal values of ALT, AST, total bilirubin, TSH, free T4, and total T3 are exclusionary regardless of any clinical significance assessment by the Investigator (see Exclusion Criteria 1 and 2).
23. Clinically significant abnormal vital signs (evaluated in the supine position after 5 minutes of rest), confirmed with retesting after at least 5 minutes of additional rest and at the discretion of the PI. Vital sign reference ranges to assess eligibility are as follows:

    1. Systolic blood pressure: >90 to ≤140 mmHg
    2. Diastolic blood pressure: ≥45 to ≤90 mmHg
    3. Pulse rate: ≥40 to ≤100 beats per minute
24. Physical examination findings that are considered clinically significant in the opinion of the Investigator and likely to adversely impact study conduct and/or interpretation are exclusionary.
25. Subjects who had major surgery (e.g., requiring general anesthesia) within 12 weeks before enrollment, or will not have fully recovered from surgery, or have surgery planned during the time the subject is expected to participate in the study, or within 4 weeks after the last dose of study drug.
26. Subjects with renal dysfunction [e.g., estimated creatinine clearance <80 mL/min/1.73 m2 at screening, calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula]. CKD-EPI should not be corrected for subjects of African ancestry.
27. Subject is an employee of the Sponsor, the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, as well as family members of the employees or the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve [AUC] | 23 days
  Pharmacokinetic parameters of atorvastatin and applicable metabolites
Time to maximum plasma concentration [Tmax] | 23 days
  Pharmacokinetic parameters of atorvastatin and applicable metabolites
Maximum plasma concentration [Cmax] | 23 days
  Pharmacokinetic parameters of atorvastatin and applicable metabolites
Minimum plasma concentration [Cmin] | 23 days
  Pharmacokinetic parameters of atorvastatin and applicable metabolites
C0 [predose] | 23 days
  Pharmacokinetic parameters of atorvastatin and applicable metabolites
Half-life [t1/2] | 23 days
  Pharmacokinetic parameters of atorvastatin and applicable metabolites
Area under the concentration time curve [AUC] | 22 days
  Pharmacokinetic parameters of rosuvastatin and applicable metabolites
Time to maximum plasma concentration [Tmax] | 22 days
  Pharmacokinetic parameters of rosuvastatin and applicable metabolites
Maximum plasma concentration [Cmax] | 22 days
  Pharmacokinetic parameters of rosuvastatin and applicable metabolites
Minimum plasma concentration [Cmin] | 22 days
  Pharmacokinetic parameters of rosuvastatin and applicable metabolites
C0 [predose] | 22 days
  Pharmacokinetic parameters of rosuvastatin and applicable metabolites
Half-life [t1/2] | 22 days
  Pharmacokinetic parameters of rosuvastatin and applicable metabolites

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 23 days for part 1
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 22 days for part 2
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Time to maximum plasma concentration [Cmax] of ALG-055009 (ng/mL) | up to 23 days for part 1
  Pharmacokinetic parameters of ALG-055009 and applicable metabolites
Minimum plasma concentration [Cmin] of ALG-055009 (ng/mL) | up to 23 days for part 1
  Pharmacokinetic parameters of ALG-055009 and applicable
Area under the concentration time curve [AUC] of ALG-055009 (ng/mL)PK | up to 23 days for part 1
  Pharmacokinetic parameters of ALG-055009 and applicable metabolites
Time to maximum plasma concentration [Tmax] of ALG-055009 (ng/mL) | up to 23 days for part 1
  Pharmacokinetic parameters of ALG-055009 and applicable metabolites
Half-life [t1/2] of ALG-055009 (ng/mL) | up to 23 days for part 1
  Pharmacokinetic parameters of ALG-055009 and applicable metabolites
Time to maximum plasma concentration [Cmax] of 2-hydroxy-atorvastatin (ng/mL) | up to 23 days for part 1
  Pharmacokinetic parameters of 2-hydroxy-atorvastatin and applicable
Minimum plasma concentration [Cmin] of 2-hydroxy-atorvastatin (ng/mL) | up to 23 days for part 1
  Pharmacokinetic parameters of 2-hydroxy-atorvastatin and applicable metabolites
Area under the concentration time curve [AUC] of 2-hydroxy-atorvastatin (ng/mL) | up to 23 days for part 1
  Pharmacokinetic parameters of atorvastatin and applicable metabolites
Time to maximum plasma concentration [Tmax] of 2-hydroxy-atorvastatin (ng/mL) | up to 23 days for part 1
  Pharmacokinetic parameters of 2-hydroxy-atorvastatin and applicable metabolites
Half-life [t1/2] of 2-hydroxy-atorvastatin (ng/mL) | up to 23 days for part 1
  Time to maximum plasma concentration [Cmax] of ALG-055009 (ng/mL)
Minimum plasma concentration [Cmin] of ALG-055009 (ng/mL) | up to 22 days for part 2
  Pharmacokinetic parameters of ALG-055009 and applicable metabolites
Area under the concentration time curve [AUC] of ALG-055009 (ng/mL) | up to 22 days for part 2
  Pharmacokinetic parameters of ALG-055009 and applicable metabolites
Time to maximum plasma concentration [Tmax] of ALG-055009 (ng/mL) | up to 22 days for part 2
  Pharmacokinetic parameters of ALG-055009 and applicable metabolites
Half-life [t1/2] of ALG-055009 (ng/mL) | up to 22 days for part 2
  Pharmacokinetic parameters of ALG-055009 and applicable metabolites
Time to maximum plasma concentration [Cmax] of rosuvastatin (ng/mL) | up to 22 days for part 2
  Pharmacokinetic parameters of rosuvastatin and applicable metabolites
Minimum plasma concentration [Cmin] of rosuvastatin (ng/mL) | up to 22 days for part 2
  Pharmacokinetic parameters of rosuvastatin and applicable metabolites
Area under the concentration time curve [AUC] of rosuvastatin (ng/mL) | up to 22 days for part 2
  Pharmacokinetic parameters of rosuvastatin and applicable metabolites
Time to maximum plasma concentration [Tmax] of rosuvastatin (ng/mL | up to 22 days for part 2
  Pharmacokinetic parameters of rosuvastatin and applicable metabolites
Half-life [t1/2] of rosuvastatin (ng/mL) | up to 22 days for part 2
  Pharmacokinetic parameters of rosuvastatin and applicable metabolites

OTHER OUTCOMES:
Cholesterol | up to 23 days for part 1
  Monitor plasma cholesterol and 4β-OH-cholesterol levels as a potential CYP3A4 induction marker
Cholesterol | Up to 22 days for part 1
  Monitor plasma cholesterol and 4β-OH-cholesterol levels as a potential CYP3A4 induction marker

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Austin Research Unit, Austin, Texas, United States